CLINICAL TRIAL: NCT05202470
Title: Effectiveness of Telehealth Program in Patients With Type 2 Diabetes: Randomized Controlled Study
Brief Title: Effectiveness of Telehealth Program in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mugla Sıtkı Kocman
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Education (TE) (Experimental): After the first meeting, diabetes education videos prepared in two parts a week will be sent to the mobile phones of the individuals. The video submission will be completed in a total of four weeks.
  Interventions: Other: TE
- Conventional Education (CE) (Active Comparator): Paper-based education forms will be given to the patients in the first group. Face-to-face conventional diabetes education will be carried out.
  Interventions: Other: CE

INTERVENTIONS:
Other: TE — After the first meeting, diabetes education videos prepared in two parts a week will be sent to the mobile phones of the individuals. The video submission will be completed in a total of four weeks.
  Arms: Telehealth Education (TE)
Other: CE — After the first meeting, diabetes education videos prepared in two parts a week will be sent to the mobile phones of the individuals. The video submission will be completed in a total of four weeks.
  Arms: Conventional Education (CE)

SUMMARY:
Diabetes education is of great importance in the effective management of diabetes. Studies have shown that patients given diabetes education have positive developments in their ability to manage the disease and their attitudes towards the disease. The aim of the study is to compare the education given to individuals with Type 2 diabetes via mobile phone and the education given to individuals via brochures with conventional methods.

DETAILED DESCRIPTION:
The use of telehealth technologies in the field of health is becoming more and more widespread. Telehealth has become one of the frequently used options in the follow-up process of chronic diseases such as diabetes, especially in recent years. Diabetes education is of great importance in the effective management of diabetes. Studies have shown that patients given diabetes education have positive developments in their ability to manage the disease and their attitudes towards the disease. The aim of the study is to compare the education given to individuals with Type 2 diabetes via mobile phone and the education given to individuals via brochures with conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of type 2 diabetes mellitus for at least 6 months,
* Those between the ages of 18-65,
* Receiving oral antidiabetic and/or insulin therapy,
* Having a mobile phone capable of receiving and playing video messages,
* Does not have hearing, speech and psychiatric problems that prevent communication,

Exclusion Criteria:

* Individuals who do not volunteered to participate in the study
* Patients who have hearing, speech and psychiatric problems that prevent communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
International Survey of Physical Activity (IPAQ) | 4 weeks
  Physical activity assessment
Goal orientation in exercise measure (GOEM) | 4 weeks
  Measurement of goal orientation in exercise
Mini Nutritional Assessment | 4 weeks
  To evaluate the nutrition status of the patients
The Problem Areas in Diabetes Scale (PADS) | 4 weeks
  PADS evaluates comprehensive diabetes evaluation. A total score is ranged between 0 - 100. Patients scoring 40 or higher may be at the level of "emotional burnout" and warrant special attention.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Tuna, PhD, Study Chair — Muğla Sıtkı Koçman University; Emine Neşe Yeniçeri, MD, Principal Investigator — Muğla Sıtkı Koçman University; Cem Şahin, MD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No